CLINICAL TRIAL: NCT04479137
Title: Possible Predictors of Mortality Based on COVID-19 for Patients Under 50 Years Old: A Multi-Center Experience of Istanbul
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ramazan Guven, Professor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KSSEAH--PPC
Record Dates: First submitted 2020-07-18; First posted 2020-07-21 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Covid-19; Risk Factor, Mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCR for COVID-19 — Novel Coronavirus 2019 DNA will be analyzed by PCR in nasopharyngeal swab

SUMMARY:
COVID-19, which emerged in China in December 2019, has become a pandemic with its spread to many countries of the world. Mortality rates of COVID-19 pandemics vary between countries. It is known that mortality based on COVID-19 is higher in old population. Therefore the aim of this study to analyze the experience of 7 governmental hospitals in terms of patient characteristics, possible risk factors of mortality based on COVID-19.

DETAILED DESCRIPTION:
COVID-19, which emerged in China in December 2019, has become a pandemic with its spread to many countries of the world. Mortality rates of COVID-19 pandemics vary between countries. It is known that mortality based on COVID-19 is higher in old population. Although several factors defined to be effective on this 'age depending factors' regional differences should be assessed deeply to clarify both the etiology and epidemiology. Therefore the aim of this study to analyze the experience of 7 governmental hospitals in terms of patient characteristics, possible risk factors of mortality based on COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* accepted to participate
* patients who were proven to have COVID-19

Exclusion Criteria:

* declined to participate
* patients whose age under 18 or more than 50 years

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Patients who were between 18-50 years of age and were died caused by COVID-19 will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
mortality based on COVID-19 | 3 months
  mortality based on COVID-19 within the patients aged between 18-50 will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No